CLINICAL TRIAL: NCT01615913
Title: Optimizing the Treatment of Toenail Onychomycosis Using a New Transdermal Patch Combined With Terbinafine and Ketoconazole Formulation
Brief Title: Optimizing the Treatment of Toenail Onychomycosis Using a New Transdermal Patch Combined With Terbinafine/Ketoconazole
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiwan Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TE9512
Record Dates: First submitted 2012-06-04; First posted 2012-06-11 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Onychomycosis
Keywords: onychomycosis; terbinafine; ketoconazole; transdermal topical therapy
MeSH Terms: conditions — Onychomycosis | interventions — Terbinafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3% terbinafine patch (Experimental): A 10-cm2 patch containing 3 mg terbinafine and 2 mg ketoconazole
  Interventions: Drug: 3 mg terbinafine and 2 mg ketoconazole containing patch
- 6% terbinafine patch (Experimental): A 10-cm2 patch containing 6 mg terbinafine and 2 mg ketoconazole
  Interventions: Drug: 6 mg terbinafine and 2 mg ketoconazole containing patch
- 8% terbinafine patch (Experimental): A 10-cm2 patch containing 8 mg terbinafine and 2 mg ketoconazole
  Interventions: Drug: 8 mg terbinafine and 2 mg ketoconazole containing patch

INTERVENTIONS:
Drug: 3 mg terbinafine and 2 mg ketoconazole containing patch — A novel transdermal patch that is to be used to treat toenail onychomycosis with minimal body exposure to the antifungal drugs. The active substances in the patch are 3% terbinafine (contains 3-mg terbinafine/patch) and 2% ketoconazole (contains 2-mg ketoconazole/patch). The average daily released drug amount estimated from in-vitro skin permeation test were about 3.99 mcg for terbinafine and 1.70 mcg for ketoconazole, respectively.
  Arms: 3% terbinafine patch
Drug: 6 mg terbinafine and 2 mg ketoconazole containing patch — A novel transdermal patch that is to be used to treat toenail onychomycosis with minimal body exposure to the antifungal drugs. The active substances in the patch are 6% terbinafine (contains 6-mg terbinafine/patch) and 2% ketoconazole (contains 2-mg ketoconazole/patch). The average daily released drug amount estimated from in-vitro skin permeation test were about 8.52 mcg for terbinafine and 2.03 mcg for ketoconazole, respectively.
  Arms: 6% terbinafine patch
Drug: 8 mg terbinafine and 2 mg ketoconazole containing patch — A novel transdermal patch that is to be used to treat toenail onychomycosis with minimal body exposure to the antifungal drugs. The active substances in the patch are 8% terbinafine (contains 8-mg terbinafine/patch) and 2% ketoconazole (contains 2-mg ketoconazole/patch). The average daily released drug amount estimated from in-vitro skin permeation test were about 10.7 mcg for terbinafine and 2.17 mcg for ketoconazole, respectively.
  Arms: 8% terbinafine patch

SUMMARY:
This study is to explore the optimization of anti-onychomycosis patch with various formulation contents (three patch groups: 3%, 6% and 8% of terbinafine (contains 3-mg, 6-mg and 8-mg/patch terbinafine, respectively) combined with fixed 2% ketoconazole (contains 2-mg ketoconazole/patch) and its safety profile.

DETAILED DESCRIPTION:
This study is to explore the optimization of anti-onychomycosis patch with various formulation contents (three patch groups: 3%, 6% and 8% of terbinafine (contains 3-mg, 6-mg and 8-mg/patch terbinafine, respectively) combined with fixed 2% ketoconazole (contains 2-mg ketoconazole/patch) and its safety profile. At least 18 patients (age: 20 to 75 years old) with one or two feet toenails infected simultaneously need to complete the whole study. Patients will be assigned to one of patch groups. The patients with only one infected toenail will also apply one patch on other foot with uninfected toenail. The patch will be applied on the foot on the dorsal site and leave it there for two consecutive days. Totally six patches will be used for each week. The duration of therapy will be 24 weeks. The patients' blood sample and toenail clippings will be collected every 8 weeks and will be analyzed as well as the safety profiles. The most appropriate patch formulation will be selected on the drug content residues in toenail. The safety profile will be also presented and discussed with various anti-onychomycosis patch formulations.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 20-75 years of age
* Fungal infection of one or both toenails will be confirmed using the method of histopathological examination with periodic acid-Schiff (PAS) staining (Yang JH, et al., 2007)
* The toenail infection can be due to a dermatophyte, yeast or mixed infections (dermatophyte and non-dermatophyte)
* The target toenail area must have at least 25% to no more than 75% disease involvement without spikes
* Patients agree to sign the informed consent form

Exclusion Criteria:

* Using any kind of systemic or topical nail lacquer solution antifungal drugs within 6 months before at screening visit; or using any other topical antifungal agents, such as ointment, cream, gel, solution, suspension, oil or lotion forms, within two weeks before at screening visits
* Patients with the target toenail involving the matrix (lunula) or having less than 2 mm clear (unaffected) nail plate length beyond the proximal fold
* Presence of dermatophytoma on the target nail
* Using professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit
* Patients who are unwilling to provide nail clippings
* Patients who have been previously reported to be allergic to topical or systemic terbinafine or ketoconazole therapy or both
* Known pregnancy or plan to get pregnant within study duration or lactation at time of enrollment
* Unconsciousness or inability to understand this form or this study project.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Presented by pharmacokinetic data (drug plasma concentrations vs. time) or drug deposit amounts in feet nails. | baseline, 8-week, 16-week and 24-week
  Both terbinafine and ketoconazole plasma concentration, and their residual contents in toenails will be measured with a validated LC/MS-MS method.

SECONDARY OUTCOMES:
(1) Efficacy is evaluated 24 weeks after the start of treatment and will be recorded at baseline, 8-week, 16-week and 24-week. | baseline, 8-week, 16-week and 24-week
  The degrees of improvement are assessed based on each toenail as follows:
  1. Complete cure is defined as regeneration of a healthy nail plate to replace the diseased nail.
  2. Marked improvement is defined as regeneration of a healthy nail plate in at least 70% of the affected nail.
  3. Improvement is defined as regeneration in 40-70% of the affected nail.
  4. Slight improvement is defined as regeneration in less than 40%.
  5. No change is defined as the absence of change or exacerbation of the disease condition or the side effect.
(2) Safety Monitoring | baseline, 8-week, 16-week and 24-week
  Adverse events, both local and systemic, will be recorded and their relation to the trial drugs is judged.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan, Taiwan